CLINICAL TRIAL: NCT00230490
Title: Open-label Treatment Extension Study for Patients Who Complete Study RNA200103-201
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Adverse findings from nonclinical carcinogenicity studies.
Sponsor: Bausch Health Americas, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RNA200103-202
Record Dates: First submitted 2005-09-28; First posted 2005-09-30 (Estimated); Last update posted 2019-11-29 (Actual); Status verified 2019-11

CONDITIONS: Hepatitis B, Chronic
Keywords: Hepatitis B, Chronic; Hepatitis B Virus; Pradefovir Mesylate; Adefovir Dipivoxyl
MeSH Terms: conditions — Hepatitis B, Chronic; Hepatitis B | interventions — pradefovir

INTERVENTIONS:
Drug: pradefovir mesylate
Drug: adefovir dipivoxyl

SUMMARY:
Compare the long-term safety of pradefovir to adefovir dipivoxyl

DETAILED DESCRIPTION:
* Compare the long-term safety of pradefovir to adefovir dipivoxyl
* Monitor development of resistance
* Evaluate virologic and biochemical response

ELIGIBILITY:
Inclusion Criteria:

* Patients who completed 48 weeks of treatment in study RNA200103-201

Exclusion Criteria:

* Patients who were determined to be treatment failures in study RNA200103-201
* Patients who experienced a serious adverse event judged to be related to study drug in study RNA200103-201
* Patients with a serum creatinine greater than 2.0 mg/dl on two consecutive determinations in study RNA200103-201

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 150
Dates: Start 2005-06; Study Completion 2007-05 (Actual)

PRIMARY OUTCOMES:
- Safety: Clinical examinations of laboratory tests
- Efficacy: Change in viral load over time

SECONDARY OUTCOMES:
- Efficacy: Proportion of patients with undetectable viral load

CONTACTS AND LOCATIONS:
Overall Officials: Ralph T. Doyle, Study Director — Bausch Health Americas, Inc.